CLINICAL TRIAL: NCT05670496
Title: Collection of Clinical Data and Specimens for Research in Hearing, Balance, Taste, Smell, Voice, Speech, and Language Disorders.
Status: Recruiting | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001126; 001126-DC
Record Dates: First submitted 2022-12-31; First posted 2023-01-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Hearing Loss; Deafness
Keywords: Deafness; Hearing; Speech; Vestibular; Audiology; Natural History
MeSH Terms: conditions — Hearing Loss; Deafness; Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients at risk, suspected of having, have a history of, or currently have a diagnosed hearing, balance or communication disorder.

SUMMARY:
Background:

People with hearing, balance, and taste, smell, voice, speech, language, and other Ear, Nose, and Throat (ENT) disorders may seek treatment at the National Institute on Deafness and Other Communication Disorders (NIDCD). Some of these people may benefit from enrolling in the NIDCD intramural research program to receive their care. Enrolling will also allow investigators to collect participants clinical data and specimens for future research.

Objective:

This natural history study has 2 goals: (1) to collect data and specimens that may be used for research; and (2) to evaluate participants who may be candidates for other research studies.

Eligibility:

People aged 2 years or older with a hearing, balance, and communication disorder. Those at risk or who are suspected of having such a disorder are also eligible.

Design:

Participants will be screened. Their medical records will be reviewed.

Participants will agree to have their medical data used for research. Specimens such as blood or other tissue samples may also be used for research. All data and specimens will be collected during their routine care visits.

All tests done will be the normal care for each participant s condition. No tests will be done solely for research.

Some of these tests may require blood or tissue samples. Some may use special tools to test hearing and balance. Some may test heart or lung function. These tests may also include different types of imaging scans.

All tests will be explained. Participants may ask questions at any time.

Participants may remain in this study for up to 2 years. If they need further care, they may sign a new consent.

...

DETAILED DESCRIPTION:
Study Description:

It may be in the interest of the NIDCD Clinical Research Program (CRP) to collect clinical data or specimens generated in the diagnosis and treatment of hearing, balance, taste, smell, voice, speech, language, and other Ear, Nose, and Throat (ENT) disorders and to evaluate patients to determine candidacy for intramural clinical studies. This protocol will provide the administrative vehicle to enable the evaluation and provision of clinical care for patients with hearing, balance and communication disorders by the NIDCD CRP, Clinical Center, and consult services as well as to provide a repository of information on enrolled subjects to allow for hypothesis generation in future research. No investigational therapies will be administered in this study. As part of hypothesisgenerating research related to taste and oral sensation, participants may undergo brief sensory testing using food-grade tannic acid solutions. This testing is designed to characterize taste, mouthfeel, and chemesthetic responses and does not involve administration of investigational agents or swallowing of test solutions.

Objectives:

* To provide a repository of data and samples collected from clinical data or specimens generated in the diagnosis and treatment of hearing, balance, taste, smell, voice, speech, language, and other ENT disorders to allow for hypothesis generation in future research.
* To evaluate patients to determine candidacy for intramural clinical studies

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Patients must be age 2 years or older if procedures or treatment are required.
* Patients at risk, suspected of having, have a history of, or currently have a diagnosed hearing, balance, taste, smell, voice, speech, language, and other ENT disorder.
* An NIDCD clinical investigator and PI determines it is in the interest of the patient/individual and NIDCD CRP for the subject to undergo consult, treatment or follow-up at the NIDCD/NIH
* Patient or their Legally Authorized Representative is able to provide informed consent. The consent form will be signed by parents or guardians of patients under the age of 18.
* A subset of enrolled participants with known or suspected PIEZO2-related sensory dysfunction may be asked to participate in the remote taste and oral somatosensory testing procedures. Participation in this component is optional and not required for enrollment or continued participation in the parent protocol.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Candidates who do not meet the inclusion criteria.
* Candidates who in the opinion of the PI and clinical team have medical or unstable conditions for which NIDCD and CC consultative services are unable to provide or support optimal care

Participants without known or suspected PIEZO2-related sensory dysfunction will not be asked to complete the sensory testing component. Additional exclusion criteria for taste testing only procedures include:

* Active oral sores, open cuts, or significant oral pain
* Recent oral surgery or dental procedures within the past 7 days
* Known allergy or hypersensitivity to tannins or polyphenols
* Acute upper respiratory infection or conditions that may interfere with taste perception

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at risk, suspected of having, have a history of, or currently have a diagnosed hearing, balance and communication disorders referred to NIDCD Clinical Investigators by the Intramural Consult Service or community providers
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical data collection | Ongoing
  To collect clinical data or specimens generated in the diagnosis and treatment of hearing, balance and communication disorders
Evaluation for clinical studies | Ongoing
  To evaluate patients to determine candidacy for intramural clinical studies

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Levy, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001126-DC.html